CLINICAL TRIAL: NCT01188031
Title: A Relative Bioavailability Study of 2 mg Alprazolam Oral Disintegrating Tablets Under Fasting Conditions
Brief Title: A Relative Bioavailability Study of 2 mg Alprazolam OD Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Meena Venugopal, Director, Clinical R&D, Actavis Inc
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: R06-0302
Record Dates: First submitted 2010-08-23; First posted 2010-08-25 (Estimated); Last update posted 2010-08-25 (Estimated); Status verified 2010-08

CONDITIONS: Healthy
Keywords: Bioequivalence; ALPRAZOLAM; Healthy subjects
MeSH Terms: interventions — Alprazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ALPRAZOLAM ORALLY DISINTEGRATING TABLETS (Experimental): ALPRAZOLAM ORALLY DISINTEGRATING TABLETS, 2.0 MG, single dose
  Interventions: Drug: ALPRAZOLAM ORALLY DISINTEGRATING TABLETS, 2.0 MG
- NIRAVAM TM (Active Comparator): NIRAVAM TM 2 mg orally disintegrating tablets, single dose
  Interventions: Drug: NIRAVAM TM 2 mg orally disintegrating tablets, single dose

INTERVENTIONS:
Drug: ALPRAZOLAM ORALLY DISINTEGRATING TABLETS, 2.0 MG — A: Experimental Subjects received Purepac Pharmaceutical Co. formulated products under fasting conditions
  Other Names: NIRAVAM
  Arms: ALPRAZOLAM ORALLY DISINTEGRATING TABLETS
Drug: NIRAVAM TM 2 mg orally disintegrating tablets, single dose — B: Active comparator Subjects received Schwarz Pharma Inc. formulated products under fasting conditions
  Other Names: ALPRAZOLAM
  Arms: NIRAVAM TM

SUMMARY:
This study compared the relative bioavailability (rate and extent ofbsorption) of Alprazolam Orally Disintegrating Tablets, 2.0 mg by Purepac Pharmaceutical Co. with that of Niravam' 2 mg Orally Disintegrating Tablets manufactured for Schwarz Pharma, Inc. (by Cima Labs Inc.®)following a single, oral dose (I x 2 mg disintegrating tablet) in healthy adult volunteers administered under fasting conditions.

DETAILED DESCRIPTION:
Study Type: Interventional Study Design: This was a single-center, randomized, two-way crossover study conducted under fasting conditions Official Title: A Relative Bioavailability Study of 2 mg Alprazolam Oral Disintegrating Tablets under Fasting Conditions

Further study details as provided by Actavis Elizabeth LLC:

Primary Outcome Measures:

Rate and Extend of Absorption

ELIGIBILITY:
Inclusion Criteria:

Subjects who met the following criteria were included in the study.

1. Volunteers who were informed of the nature of the study and who read, reviewed, and signed the informed consent prior to Period I dosing.
2. Volunteers who completed the screening process within 28 days prior to Period I dosing.
3. Volunteers who were healthy adult men and women 18 years of age or older at the time of dosing.
4. Volunteers who had a body mass index (BMI) between 18-32 kg/nr', inclusive, and weighed at least 110 lbs.
5. Volunteers who were healthy as documented by the medical history, physical examination (including but may not be limited to an evaluation of the cardiovascular, gastrointestinal, respiratory and central nervous systems), vital sign assessments, 12-lead electrocardiogram (ECG), clinical laboratory assessments, and by general observations. Any abnormalities/deviations form the normal range that were considered clinically relevant by the study physician and investigator were evaluated for individual cases, documented in study files, and agreed upon by both the study physician and investigator prior to enrolling the volunteer in this study and for continued enrollment.
6. Female volunteers ofpostmenopausal (no menses) status for at least 1 year and has a serum FSH level 2: 30 mlU/mL or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy.)

Exclusion Criteria:

Subjects who met any ofthe following criteria were excluded from the study.

1. Volunteers who reported receiving any investigational drug within 28 days prior to Period I dosing.
2. Volunteers who reported any presence or history of a clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine, or neurologic system(s) or psychiatric disease as determined by the clinical investigator(s).
3. Volunteers whose clinical laboratory test values outside the accepted reference range and, when confirmed on re-examination, were deemed clinically significant.
4. Volunteers who demonstrated a reactive screen for hepatitis B surface antigen, hepatitis C antibody, or HIV antibody.
5. Volunteers who reported a history of allergic response(s) to alprazolam or related drugs.
6. Volunteers who reported the use of any systemic prescription medication in the 14 days prior to Period I dosing.
7. Volunteers who reported the use of any drug known to induce or inhibit hepatic drug metabolism in the 28 days prior to Period I dosing.
8. Volunteers who reported a history ofclinically significant allergies including drug allergies.
9. Volunteers who reported a clinically significant illness during the 4 weeks prior to Period I dosing (as determined by the clinical investigators).
10. Volunteers who reported a history of drug or alcohol abuse addiction or abuse within the past year.
11. Volunteers who demonstrated a positive drug abuse screen for this study prior to Period I dose administration.
12. Volunteers who currently used tobacco products.
13. Volunteers who reported donating greater than 150 mL ofblood within 28 days prior to Period I dosing. All subjects were advised not to donate blood for four weeks after completing the study.
14. Volunteers who donated plasma (e.g. plasmapheresis) within 14 days prior to Period I dosing. All subjects were advised not to donate plasma for four weeks after completing the study
15. Volunteers who demonstrated a positive pregnancy screen (females only).
16. Volunteers who were currently pregnant or breastfeeding (females only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-06; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Rate and Extend of Absorption | 72hr

CONTACTS AND LOCATIONS:
Overall Officials: James D. Carlson,, Pharm.D,, Principal Investigator — PRACS Institute, Ltd.
Locations (1):
- PRACS Institute, Ltd., Fargo, North Dakota, United States